CLINICAL TRIAL: NCT05457036
Title: Evaluation of the Effect of Spry Belt Treatment on Bone Turnover Marker Profile in a 12-week, Sham-controlled Clinical Study
Brief Title: Evaluation of the Effect of Spry Belt Treatment on Bone Turnover Marker Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bone Health Technologies, Inc. (Industry)
Collaborators: University of Nebraska (Other); University of California, San Francisco (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRD-09-1471; SB1AG046005 (NIH)
Record Dates: First submitted 2022-07-09; First posted 2022-07-13 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Osteopenia; Low Bone Density
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: After signing the Study consent form, the subject will be randomized (1:1, block randomization with a block size of 10 stratified by site and race (Caucasian or non-Caucasian)) to one treatment group (Active or Sham treatment, see below) and be considered part of the intent-to-treat (ITT) cohort.
Who Masked: Participant, Care Provider
Masking Description: Research staff will not change any study procedures based on the subject's group placement. Blinding assessment will be done during the study visits 2 and 3. We will use an established blinding assessment.33 Subjects will be asked if they believe they are receiving the real treatment, sham/placebo treatment, or if they are uncertain. Answers will be asked and recorded by the research staff on the case report forms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Treatment Group (Experimental): Active Treatment device device provides gentle energy to the lower spine and hips.
  Interventions: Device: Spry Belt
- Sham Treatment Group (Sham Comparator): Sham Treatment device is identical to the Active Treatment device except the sham device does not produce the gentle energy.
  Interventions: Device: Sham Spry Belt

INTERVENTIONS:
Device: Spry Belt — The Spry Belt is a device worn around the hips which delivers gentle energy to the lower back. The level of energy is controlled by an internal microprocessor (computer) so that it is safe and comfortable. The energy is at a level that may or may not be perceptible to the user. The device is powered by an internal lithium-ion battery which must be recharged periodically. The device is designed to be used with its companion Spry app (via Bluetooth Low Energy (BLE)) so that anonymous usage statistics may be monitored. The expected shelf life of the device is longer than 2 years and the expected use life is at least 12-18 months.
  Arms: Active Treatment Group
Device: Sham Spry Belt — The Sham Spry Belt is a device worn around the hips which does not deliver gentle energy to the lower back. The device instead provides a clicking noise similar to a motor. The device is powered by an internal lithium-ion battery which must be recharged periodically. The device is designed to be used with its companion Spry app (via BLE) so that anonymous usage statistics may be monitored. The expected shelf life of the device is longer than 2 years and the expected use life is at least 12-18 months.
  Arms: Sham Treatment Group

SUMMARY:
To conduct a sham-controlled study to rigorously evaluate the effect of Spry Belt treatment on key bone turnover markers (BTMs) over a 12-week period. The investigators will calculate the percentage and absolute changes from baseline for several BTMs for both the active and sham treatment groups.

DETAILED DESCRIPTION:
This will be a 12-week, randomized, controlled study with 90 subjects. At enrollment, subjects will be randomized to the Active Treatment or Sham Treatment. All subjects will receive dietary supplements (calcium and vitamin D) for the duration of the study. Subjects will be asked to self-administer daily at-home treatments with the device at least 5 times each week. The investigators will evaluate safety via adverse events reported to the research staff and via responses to a survey on potential side effects. DXA scans will be obtained at the Screening Visit and Visit 3 (Study Completion). Blood and urine will be collected at Day 0 (Visit 1), Week 6 (Visit 2), and Week 12 (Visit 3).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Had her last menstrual period at least one year prior to the time of study enrollment
* Has low bone mass as defined by a DXA T-score between -1.0 and -2.49 for the femoral neck, total femur, or lumbar spine
* Is 50 years of age or older
* Can walk and stand without an assistive device
* Is able to provide informed consent
* Is able to understand spoken and written English
* Is capable and willing to follow all study-related procedures

Exclusion Criteria:

* Has a bone mineral density (BMD) at the femoral neck, total femur, or lumbar spine of T score ≤ -2.5 (defined by DXA)
* Has a 10-year probability of major fracture >20% or hip fracture >3% based on results of the Fracture Risk Assessment (FRAX) Tool (at screening)
* Is currently taking or has taken oral bisphosphonates or other prescription osteoporosis medications in the past 24 months, or estrogen replacement therapy, glucocorticosteroids, dehydroepiandrosterone, tenofovir disoproxil fumarate, or other drugs affecting bone in the past 3 months
* Has had at least one fracture or at least one major surgery within the past 6 months
* Smokes >10 cigarettes per day over the past 6 months
* Has had an average of 14 alcoholic drinks per week over the past 6 months
* Has type I diabetes
* Has a history of severe renal disease or kidney failure
* Has had bariatric surgery
* Has been diagnosed with chronic renal disease, cirrhosis, multiple myeloma, neuromuscular disease, osteomalacia, Paget's disease, osteogenesis imperfecta, severe osteoarthritis, rheumatoid arthritis, severe peripheral neuropathy, gastrointestinal malabsorption or sprue, an eating disorder (e.g., anorexia nervosa, bulimia), uncontrolled hypertension, or chronic diseases known to affect the musculoskeletal system (e.g., muscular dystrophy)
* Has been diagnosed with an endocrine disorder known to adversely affect bone density, such as primary hyperparathyroidism, hyperthyroidism, or Cushing's syndrome, unless definitively treated
* Has cancer and/or is being treated for cancer
* Has had a bilateral oophorectomy
* Is being treated for a herniated disc
* Has had any prolonged immobilization (i.e., bedrest) for over one week or non-weight bearing for greater than one month of the axial or lower appendicular skeleton within the last 3 years
* Is engaged in high-impact activity at least three times per week (including but not limited to tennis, aerobics, running, weight-bearing activity or exercise more intense than fast walking)
* Has a known allergy to neoprene
* Has a hip circumference >56 inches
* Has a BMI >35
* Has abnormal results for the following laboratory tests:
* Serum 25(OH)D outside of the range: 10-100 ng/mL
* Serum calcium outside of the normal laboratory ranges
* Serum PTH outside of the normal laboratory ranges
* TSH outside of the normal laboratory ranges*
* FSH less than 40 (mIU/L) **
* Has joint replacement implants in the ankle, knee, or hip
* Has had a spinal fusion procedure
* Has an active implant (e.g. implanted neurostimulator) in the areas of the lumbar or thoracic spine, pelvis, or buttocks
* Has had a major change in high-impact physical activity level (increase or decrease) in the past 3 months
* Has undergone or is undergoing transgender hormone therapy
* Is deemed unsuitable for enrollment in the study by the Principal Investigator

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female who had her last menstrual period at least one year prior to the time of study enrollment
Enrollment: 94 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline for Urinary N-telopeptide (uNTX) | 6 weeks
  The percent change from Baseline for both Active and Sham treatment groups compared with a two-sample t-test with a significance level of 0.05.
Adverse Event Safety Endpoint | 12 weeks
  Adverse Events as recorded on the Adverse Event Case Report Form, showing number and type of Serious Adverse Events and Device Related-Adverse Events compared between the Active and Sham groups

SECONDARY OUTCOMES:
Secondary Safety Endpoint | 12 weeks
  The prevalence and severity of all side effects, as measured via the Adverse Event Checklist, will be compared between the Active and Sham groups. We will perform separate sub-comparisons for side effects that subjects' report as likely to be due to Spry Belt treatment and for those that are not.
DXA-based Lumbar Spine Bone Mineral Density (aBMD) | 12 weeks
  For each subject, aBMD for the lumbar spine (L1-L4 vertebrae) will be calculated at Baseline and 12 weeks (Study Completion). The percent change in aBMD will then be calculated for each subject. Results for the Active and Sham groups will be compared using a with a two-sample t-test with a significance level of 0.05.
DXA-based Total Femur Bone Mineral Density (aBMD) | 12 weeks
  For each subject, aBMD for the total femur (average of left and right femurs) will be calculated at Baseline and 12 weeks (Study Completion). The percent change in aBMD will then be calculated for each subject. Results for the Active and Sham groups will be compared using a with a two-sample t-test with a significance level of 0.05.
Serum amino-terminal propeptide of type 1 procollagen (P1NP) | 12 weeks
  For each subject, sP1NP samples will be collected at Baseline, 6 weeks (Visit #2), and 12 weeks (Visit #3, Study Completion). The percent change in sP1NP will then be calculated for each subject.
Serum N-telopeptide (sNTX) | 12 weeks
  For each subject, sNTX samples will be collected at Baseline, 6 weeks (Visit #2), and 12 weeks (Visit #3, Study Completion). The percent change in sNTX will then be calculated for each subject.
Urine N-telopeptide (uNTX) | 12 weeks
  In addition to the primary endpoint, percent change in uNTX will be calculated for each subject from Baseline and 12 weeks (Visit #3, Study Completion).
Serum cross-linked C-telopeptide of type I collagen (sCTX) | 12 weeks
  For each subject, sCTX samples will be collected at Baseline, 6 weeks (Visit #2), and 12 weeks (Visit #3, Study Completion). The percent change in sCTX will then be calculated for each subject.
Quality of Life (QoL) | 12 weeks
  SF-12 will be used to evaluate QoL. For each subject, the SF-12 scores will be calculated at Baseline and 12 weeks (Study Completion). Change in SF-12 score for the Active and Sham groups will be compared using a with a two-sample t-test with a significance level of 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Hillstrom, Study Director — Bone Health Technologies
Locations (2):
- United States (2):
  - Northern California Institute for Research and Education (NCIRE), San Francisco, California
  - University of Nebraska Medical Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No